CLINICAL TRIAL: NCT05403502
Title: Safety Evaluation of an Advanced Hybrid Closed Loop System Using Lyumjev With the Tandem t:Slim X2 Insulin Pump With Control-IQ Technology in Adults, Adolescents and Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry); Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0009650
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Control-IQ Technology; lyumjev
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- t:slim X2 insulin pump with Control-IQ technology utilizing insulin Lyumjev® (Experimental): Current Control-IQ technology users with type 1 diabetes, age 6-80, will use the t:slim X2 insulin pump with Control-IQ technology 1.5 and Lyumjev insulin for 3-months of outpatient use.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ technology 1.5

INTERVENTIONS:
Device: t:slim X2 insulin pump with Control-IQ technology 1.5 — t:slim X2 insulin pump with Control-IQ technology 1.5, and wearing the Dexcom G6 sensor, used with Lyumjev® insulin.

SUMMARY:
Prospective, multi-center, single-arm study in adults and children ages 6 to 80 with type 1 diabetes to evaluate the safety of Lyumjev with Control-IQ technology to achieve labeling updates for Lyumjev and the t:slim X2 insulin pump.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study in adults and children (ages 6 to 80 years) with type 1 diabetes who are current users of the t:slim X2 insulin pump with Control-IQ technology to achieve labeling updates for Lyumjev and the t:slim X2 insulin pump. After a run-in period, participants will use the study pump with Control-IQ technology 1.5 and Lyumjev insulin for a 3-month outpatient treatment period. Up to 200 participants will be enrolled so at least 160 complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 to <81 years
2. Diagnosis of type 1 diabetes for at least 1 year
3. Currently using Control-IQ technology for at least 3 months, with CGM data recorded indicative of system use (active closed loop) for at least 85% of the possible time in 14 days prior to enrollment
4. Total daily insulin dose (TDD) at least 2 U/day
5. HbA1c < 10.5%
6. Residing full-time in the United States, with no anticipated travel outside the United States during the period of study participation.
7. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency, and willing to use the Dexcom Follow app (with push notifications turned on) for the duration of the study.
8. If >18 years old, participant has someone who lives within 30 minutes of them who is willing to be contacted if the study team can't reach the participant in case of a suspected medical emergency.
9. Participant has agreed to participate in the study; and has read, understood and signed the informed consent form (ICF) and assent, if applicable; and has agreed to follow all study procedures, including:

   1. suspending use of any personal CGM for the duration of the clinical trial once the study CGM is in use
   2. switching to or continuing to use Humalog during the lead-in period
   3. switching to Lyumjev for the main study period.
   4. willing and able to perform the study exercise and meal challenges.
10. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol, including ability to respond to alerts and alarms, and to provide basic diabetes self-management.
11. Participant and/or parent/legal guardian have the ability to read and understand English

Exclusion Criteria:

1. More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months
2. More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months
3. Inpatient psychiatric treatment in the past 6 months
4. History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or unwillingness to agree to abstain from illicit drugs throughout the study.
5. For Female: Currently pregnant or planning to become pregnant during the time period of study participation

   1. A negative pregnancy test will be required for all females of child-bearing potential (menarchal)
   2. Counseling on appropriate birth control options will be provided to females with child-bearing potential in the event the participant does not have an acceptable plan.
6. Adults lacking the capacity to provide consent and/or follow study procedures in the opinion of the investigator
7. Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
8. Hemophilia or any other bleeding disorder
9. Hemoglobinopathy
10. History of heart, liver, lung or kidney disease determined by investigator to interfere with the study
11. History of allergic reaction to Humalog or Lyumjev
12. Use of glucocorticoids, beta blockers or other medications determined by investigator to interfere with study
13. Abnormal screening electrocardiogram consistent with increased risk during exercise, such as arrhythmia, ischemia, or prolonged QTc interval (>450 ms) (Screening ECG only required for participants age > 50 years, duration of diabetes > 20 years, or history of coronary artery disease)
14. Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
15. History of adrenal insufficiency
16. History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
17. History of gastroparesis
18. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
19. Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for during the time period of study participation
20. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., Eli Lilly and Co., or TypeZero Technologies, LLC, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care
Locations (13):
- United States (13):
  - Children's Hospital Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Barbara Davis Center, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - Indiana University / Riley Hospital for Children, Indianapolis, Indiana
  - Iowa Diabetes and Endocrinology Research Center (IDERC), West Des Moines, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Diabetes & Glandular Disease (DGD), San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levy CJ, Bailey R, Laffel LM, Forlenza G, DiMeglio LA, Hughes MS, Brown SA, Aleppo G, Bhargava A, Shah VN, Clements MA, Kipnes M, Bruggeman B, Daniels M, Rodriguez H, Calhoun P, Lum JW, Sasson-Katchalski R, Pinsker JE, Pollom R, Beck RW; TL1 Study Group. Multicenter Evaluation of Ultra-Rapid Lispro Insulin with Control-IQ Technology in Adults, Adolescents, and Children with Type 1 Diabetes. Diabetes Technol Ther. 2024 Sep;26(9):652-660. doi: 10.1089/dia.2024.0048. Epub 2024 May 22. PMID 38696672

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 179 participants completed the Humalog run-in and initiated Lyumjev use.
Groups:
- Users of Tandem t:Slim X2 Insulin Pump With Control-IQ 1.5 Technology: Current Control-IQ technology users with type 1 diabetes, age 6-80, using the t:slim X2 insulin pump with Control-IQ technology 1.5, wearing the Dexcom G6 sensor who progressed to the Lyumjev Treatment Period after participating in the Humalog Lead-In Period.
Period: Humalog Lead-In Period
Arm/Group | Users of Tandem t:Slim X2 Insulin Pump With Control-IQ 1.5 Technology
Started | 183
Completed | 179
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 1
Period: Lyumjev Treatment Period
Arm/Group | Users of Tandem t:Slim X2 Insulin Pump With Control-IQ 1.5 Technology
Started | 179
Completed | 173
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- Users of Control-IQ 1.5 Technology Who Initiated the Lyumjev Treatment Period: Current Control-IQ technology users with type 1 diabetes, age 6-80, using the t:slim X2 insulin pump with Control-IQ technology 1.5, wearing the Dexcom G6 sensor and using Lyumjev insulin
Arm/Group | Users of Control-IQ 1.5 Technology Who Initiated the Lyumjev Treatment Period
Number analyzed (Participants) | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 109
  Between 18 and 65 years | 61
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 165
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 166
  More than one race | 4
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 179
Diabetes Duration at Enrollment [Mean (Standard Deviation); unit: years] | 14 (13)

OUTCOME MEASURES:

1. Primary Outcome: Severe Hypoglycemia
Description: Number of severe hypoglycemia events (with cognitive impairment such that assistance of another individual is needed for treatment) during study
Time Frame: 15 weeks
Measure: Number; unit: events
Groups:
- Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin: Current Control-IQ technology users with type 1 diabetes, age 6-80, using the t:slim X2 insulin pump with Control-IQ technology 1.5, wearing the Dexcom G6 sensor who performed a Humalog Lead-In Period, and then progressed to the Lyumjev Treatment Period.
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 3

2. Primary Outcome: Diabetic Ketoacidosis
Description: Number of diabetic ketoacidosis events requiring an overnight hospitalization and diagnosis by a doctor.
Time Frame: 15 weeks
Measure: Number; unit: events
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0

3. Primary Outcome: Unanticipated Adverse Device Effects
Description: Number of unanticipated adverse device effects (UADE) events
Time Frame: 15 weeks
Measure: Number; unit: events
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0

4. Secondary Outcome: Overall Percent Time Less Than 54 mg/dL
Description: CGM overall percent time less than 54 mg/dL
Time Frame: 15 Weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.27 (0.35)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.26 (0.27)

5. Secondary Outcome: Postprandial Percent Time Less Than 54 mg/dL, Through 4 Hours After Each Meal
Description: CGM postprandial percent time less than 54 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.26 (0.44)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.31 (0.37)

6. Secondary Outcome: Overall Percent Time Less Than 70 mg/dL
Description: CGM overall percent time less than 70 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 1.4 (1.3)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 1.2 (1.0)

7. Secondary Outcome: Postprandial Percent Time Less Than 70 mg/dL, Through 4 Hours After Each Meal
Description: CGM postprandial percent time less than 70 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 1.5 (1.5)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 1.6 (1.4)

8. Other Pre Specified Outcome: Overall Percent Time in Range Between 70-180 mg/dL
Description: Overall CGM percent time in range between 70-180 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 65 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 67 (13)

9. Other Pre Specified Outcome: Percent Time in Range Between 70-180 mg/dL, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM percent time in range between 70-180 mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 62 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 64 (14)

10. Other Pre Specified Outcome: Percent Time in Range Between 70-180 mg/dL, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM percent time in range between 70-180 mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 72 (18)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 75 (15)

11. Other Pre Specified Outcome: Overall Percent Time in Range Between 70-140 mg/dL
Description: Overall CGM percent time in range between 70-140 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 40 (14)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 42 (13)

12. Other Pre Specified Outcome: Percent Time in Range Between 70-140 mg/dL, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM percent time in range between 70-140 mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 38 (14)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 40 (13)

13. Other Pre Specified Outcome: Percent Time in Range Between 70-140 mg/dL, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM percent time in range between 70-140 mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 47 (20)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 49 (18)

14. Other Pre Specified Outcome: Overall Percent Time in Range Greater Than 180 mg/dL
Description: Overall CGM percent time in range greater than 180 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 34 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 32 (13)

15. Other Pre Specified Outcome: Percent Time in Range Greater Than 180 mg/dL, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM percent time in range greater than 180 mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 36 (16)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 34 (14)

16. Other Pre Specified Outcome: Percent Time in Range Greater Than 180 mg/dL, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM percent time in range greater than 180 mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 26 (18)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 24 (15)

17. Other Pre Specified Outcome: Overall Percent Time in Range Greater Than 250 mg/dL
Description: Overall CGM percent time in range greater than 250 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 12 (10)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 11 (8)

18. Other Pre Specified Outcome: Percent Time in Range Greater Than 250 mg/dL, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM percent time in range greater than 250 mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 13 (11)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 12 (10)

19. Other Pre Specified Outcome: Percent Time in Range Greater Than 250 mg/dL, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM percent time in range greater than 250 mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 9 (9)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 8 (7)

20. Other Pre Specified Outcome: Overall CGM Hyperglycemic Events Per Week
Description: Overall CGM hyperglycemic events per week, defined as 90 or more minutes greater than 300 mg/dL within a 120 minute window
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 1.8 (1.9)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 1.6 (1.6)

21. Other Pre Specified Outcome: CGM Hyperglycemic Events Per Week, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM hyperglycemic events per week, defined as 90 or more minutes greater than 300 mg/dL within 120 minute window, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 1.5 (1.8)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 1.4 (1.5)

22. Other Pre Specified Outcome: CGM Hyperglycemic Events Per Week, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM hyperglycemic events per week, defined as 90 or more minutes greater than 300 mg/dL within 120 minute window, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.4 (0.6)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.3 (0.4)

23. Other Pre Specified Outcome: Overall CGM Hypoglycemia Events Per Week
Description: Overall CGM hypoglycemia events per week defined as 15 or more consecutive minutes less than 54 mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.46 (0.75)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.49 (0.55)

24. Other Pre Specified Outcome: CGM Hypoglycemia Events Per Week, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM hypoglycemia events per week defined as 15 or more consecutive minutes less than 54 mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.32 (0.59)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.37 (0.46)

25. Other Pre Specified Outcome: CGM Hypoglycemia Events Per Week, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM hypoglycemia events per week defined as 15 or more consecutive minutes less than 54 mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: events per week
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
events per week
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 0.09 (0.24)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 0.09 (0.14)

26. Other Pre Specified Outcome: Overall Mean Glucose
Description: Overall CGM mean glucose mg/dL
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 167 (26)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 165 (23)

27. Other Pre Specified Outcome: Mean Glucose, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM mean glucose mg/dL, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 171 (27)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 168 (25)

28. Other Pre Specified Outcome: Mean Glucose, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM mean glucose mg/dL, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 157 (28)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 156 (23)

29. Other Pre Specified Outcome: Coefficient of Variation, Overall
Description: CGM measured Coefficient of Variation, Overall
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of coefficient of variation
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 36 (5)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 36 (5)

30. Other Pre Specified Outcome: Coefficient of Variation, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM measured Coefficient of Variation, daytime only (6:00 AM - 11:59 PM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of coefficient of variation
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 36 (5)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 36 (5)

31. Other Pre Specified Outcome: Coefficient of Variation, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM measured Coefficient of Variation, nighttime only (12:00 AM - 5:59 AM)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
percentage of coefficient of variation
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 32 (8)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 33 (6)

32. Other Pre Specified Outcome: Standard Deviation of All Glucose Values, Overall (24 Hour Day)
Description: CGM measured Standard Deviation of all glucose values (mg/dL), Overall ( 24 Hour Day). Standard Deviation of Mean Glucose is shown separately in Outcome 26.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 61 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 60 (14)

33. Other Pre Specified Outcome: Standard Deviation of All Glucose Values, Daytime Only (6:00 AM - 11:59 PM)
Description: CGM measured Standard Deviation of all Glucose Values (mg/dL), daytime only (6:00 AM - 11:59 PM). Standard Deviation of Mean Glucose, Daytime only, is shown separately in Outcome 27.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 62 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 61 (14)

34. Other Pre Specified Outcome: Standard Deviation of All Glucose Values, Nighttime Only (12:00 AM - 5:59 AM)
Description: CGM measured Standard Deviation of all Glucose Values (mg/dL), nighttime only (12:00 AM - 5:59 AM). Standard Deviation of Mean Glucose, Nighttime only, is shown separately in Outcome 28.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 52 (18)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 52 (15)

35. Other Pre Specified Outcome: Postprandial Percent Time in Range Between 70-180 mg/dL, Through 4 Hours After Each Meal
Description: Postprandial CGM percent time in range between 70-180 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 55 (17)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 57 (16)

36. Other Pre Specified Outcome: Postprandial Percent Time in Range Between 70-140 mg/dL, Through 4 Hours After Each Meal
Description: Postprandial CGM percent time in range between 70-140 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 32 (14)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 33 (13)

37. Other Pre Specified Outcome: Postprandial Percent Time Greater Than 180 mg/dL, Through 4 Hours After Each Meal
Description: Postprandial CGM percent time greater than 180 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 43 (18)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 42 (16)

38. Other Pre Specified Outcome: Postprandial Percent Time Greater Than 250 mg/dL, Through 4 Hours After Each Meal
Description: Postprandial CGM percent time greater than 250 mg/dL, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of time
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 16 (14)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 15 (12)

39. Other Pre Specified Outcome: Peak Postprandial Glucose, Through 4 Hours After Each Meal
Description: Peak postprandial glucose (mg/dL), through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 244 (40)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 241 (38)

40. Other Pre Specified Outcome: Postprandial Mean Glucose, Through 4 Hours After Each Meal
Description: Postprandial CGM mean glucose (mg/dL), through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 180 (32)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 177 (28)

41. Other Pre Specified Outcome: Postprandial Incremental Area Under the Glucose Curve, Through 4 Hours After Each Meal
Description: CGM postprandial incremental area under the glucose curve, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
mg*hr/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 31 (12)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 30 (8)

42. Other Pre Specified Outcome: Coefficient of Variation, Postprandial, Through 4 Hours After Each Meal
Description: CGM measured Coefficient of Variation, Postprandial, through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: percentage of coefficient of variation
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
percentage of coefficient of variation
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 36 (6)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 36 (5)

43. Other Pre Specified Outcome: Standard Deviation of All Glucose Values, Postprandial Through 4 Hours After Each Meal
Description: CGM measured Standard Deviation of all glucose values (mg/dL), Postprandial through 4 hours after each meal. Calculated as mean (SD) over all 4 hour postprandial periods throughout the study. Standard Deviation of Mean Glucose, Postprandial through 4 hours after each meal, is shown separately in Outcome 40.
Time Frame: during 4 hour postprandial period after each meal, up to 15 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 174
mg/dL
  Humalog Lead-In Period Weeks 1-2 (2 Weeks) | 64 (15)
  Lyumjev Treatment Period Weeks 3-15 (13 Weeks) | 64 (14)

44. Other Pre Specified Outcome: HbA1c Change From Baseline
Description: Change in HbA1c from End of Humalog Lead-in Period (End of Week 2) to End of Lyumjev Treatment Period (End of Week 15)
Time Frame: 13 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 172
percentage of glycated hemoglobin | -0.1 [-0.2 to 0.0]

45. Other Pre Specified Outcome: Patient Reported Outcomes: TRIM-D
Description: Patient Reported Outcomes on the Treatment Related Impact Measure-Diabetes (TRIM-D) scale. Total score measured on a scale of 0 to 100 with higher scores indicating better diabetes treatment impact. Assessed at the start of Humalog Run-In (Start of Week 1) and again at End of Lyumjev use (End of Week 15).
Time Frame: 15 weeks
Population: 3 participants did not have data at the end of the Lyumjev treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 176
score on a scale
  Start of Humalog Lead-In Period (Start of Week 1) | 74 (12)
  Lyumjev Treatment Period (End of Week 15): number analyzed (Participants) | 173
  Lyumjev Treatment Period (End of Week 15) | 80 (12)

46. Other Pre Specified Outcome: Patient Reported Outcomes: TRIM-DD
Description: Patient Reported Outcomes on the Treatment Related Impact Measure - diabetes device (TRIM-DD) scale. Measured on a scale of 0 to 100 with higher scores indicating more positive diabetes device impact. Assessed at the start of Humalog Run-In (Start of Week 1) and again at End of Lyumjev use (End of Week 15).
Time Frame: 15 weeks
Population: 4 participants did not have data at the end of the Lyumjev treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 178
score on a scale
  Start of Humalog Lead-In Period (Start of Week 1) | 82 (11)
  Lyumjev Treatment Period (End of Week 15): number analyzed (Participants) | 174
  Lyumjev Treatment Period (End of Week 15) | 86 (12)

47. Other Pre Specified Outcome: Patient Reported Outcomes: ITSQ
Description: Patient Reported Outcomes on the Insulin Treatment Satisfaction Questionnaire (ITSQ) scale. Measured on a scale of 0 to 100 with higher scores indicating better treatment satisfaction. Assessed at the start of Humalog Run-In (Start of Week 1) and again at End of Lyumjev use (End of Week 15).
Time Frame: 15 weeks
Population: 5 participants did not have data at the end of the Lyumjev treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-Loop Use With Control-IQ 1.5 and Lyumjev Insulin
Number analyzed (Participants) | 179
score on a scale
  Start of Humalog Lead-In Period (Start of Week 1) | 75 (13)
  Lyumjev Treatment Period (End of Week 15): number analyzed (Participants) | 174
  Lyumjev Treatment Period (End of Week 15) | 80 (11)

ADVERSE EVENTS:
Time Frame: 15 weeks
Description: All participants were in the same arm, first completing 2 weeks of Humalog use, and then 13 weeks of Lyumjev use with Control-IQ technology v1.5. Adverse events are noted in which treatment period the event occurred.
Groups:
- t:Slim X2 Insulin Pump With Control-IQ Technology Utilizing Insulin Lyumjev®: Current Control-IQ technology users with type 1 diabetes, age 6-80, will use the t:slim X2 insulin pump with Control-IQ technology 1.5 for ~16 day Humalog Lead-In period and Lyumjev insulin for 3-months of outpatient use.
Arm/Group | t:Slim X2 Insulin Pump With Control-IQ Technology Utilizing Insulin Lyumjev®
All-Cause Mortality (participants affected / at risk) | 0/183
Serious Adverse Events (participants affected / at risk) | 5/183
Other Adverse Events (participants affected / at risk) | 127/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t:Slim X2 Insulin Pump With Control-IQ Technology Utilizing Insulin Lyumjev® (N=183)
Other Serious Adverse Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Diagnosis of Breast Cancer in Lyumjev Treatment Period
Other Serious Adverse Event (Infections and infestations) | 1 (1) — Diagnosis of hypovolemic shock, positive strep culture in Lyumjev Treatment Period
Severe Hypoglycemia (Endocrine disorders) | 3 (3) — Requiring third party assistance associated with seizure or loss of consciousness, in Lyumjev Treatment Period
Diabetic Ketoacidosis (DKA) (Endocrine disorders) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | t:Slim X2 Insulin Pump With Control-IQ Technology Utilizing Insulin Lyumjev® (N=183)
Hyperglycemia with or without ketosis not related to the study device (Endocrine disorders) | 5 (6) — Lyumjev Treatment Period
Hyperglycemia with or without ketosis not related to the study device (Endocrine disorders) | 4 (4) — Humalog Lead-In Period
Hyperglycemia with or without ketosis related to study device (Endocrine disorders) | 32 (40) — Lyumjev Treatment Period
Hyperglycemia with or without ketosis related to study device (Endocrine disorders) | 7 (8) — Humalog Lead-In Period
Nonglycemic adverse events (General disorders) | 81 (134) — Lyumjev Treatment Period
Nonglycemic adverse events (General disorders) | 19 (21) — Humalog Lead-In Period
Nonsevere Hypoglycemia (Endocrine disorders) | 0 (0) — Humalog Lead-In Period
Nonsevere Hypoglycemia (Endocrine disorders) | 0 (0) — Lyumjev Treatment Period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT05403502/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05403502/SAP_001.pdf